CLINICAL TRIAL: NCT05857709
Title: An Observational Study to Understand the Fitness, Body Composition, Physical Activity and Sleep Patterns in People With Cystic Fibrosis on Cystic Fibrosis Transmembrane Conductance Regulator Modulator Therapy Compared to Healthy Controls
Brief Title: Fitness, Body Composition, Physical Activity and Sleep Patterns in People With Cystic Fibrosis on Modulator Therapy.
Acronym: Understand-CF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Portsmouth (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Zoe Saynor, Reader (Associate Professor) in Clinical Exercise Physiology, University of Portsmouth
Other Study IDs: 313567
Record Dates: First submitted 2023-01-23; First posted 2023-05-15 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Cystic Fibrosis
Keywords: Exercise; Modulator therapy; Peripheral muscle function; Vascular function; Body composition; Physical activity
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic fibrosis: No intervention - only assessments.
- Healthy Control: No intervention - only assessments.

SUMMARY:
Cystic fibrosis (CF) is the most common inherited condition in the United Kingdom, affecting approximately 10,837 people. It is well recognised that regular exercise is clinically important for people with CF. Exercise function measured by the maximal oxygen consumption during a cardiopulmonary exercise test is often reduced in people with CF and this has been attributed to multiple factors including, altered heart and blood vessel function, muscle function, reduced physical activity levels and poorer sleep quality.

New medicine (modulators) have become available for many people with CF. Modulators appear able to reduce sweat chloride concentrations, improve lung function and reduce the frequency of pulmonary exacerbations in people with CF. Little evidence exists to show how they may have changed the fitness and underlying mechanisms responsible for this in people with CF.

This study aims to:

1. determine the exercise function
2. determine the blood vessel function
3. determine body composition
4. determine physical activity and sleep levels in people with CF on modulator therapy compared to a healthy controls group.

DETAILED DESCRIPTION:
CF is the most common inherited condition in the United Kingdom, affecting approximately 10,837 people. CF affects the movement of salt and water across the body which leads to a thick sticky build up of mucus causing problems in the lungs and digestive system. CF also causes problems in other parts of the body for example, the heart, the blood vessels and muscles. This can impact a person with CFs' ability to exercise which can have impact prognosis, quality of life and increase the amount of times someone with CF is admitted to hospital due to a chest infection.

For many people with CF, new medicine (modulators) have lately become accessible bringing big changes to their health. Elexacaftor-tezacaftor-ivacaftor (ETI) is the most recently approved modulator for use in people with specific CF transmembrane conductance regulator gene mutations and is now the most widely used modulator therapy. So far clinical trials have largely looked at lung function, sweat chloride levels and body mass index. The wider reaching effects of modulator therapy on exercise function has not been studied. This study will see if people with CF have blood vessel and exercise dysfunction, abnormal body composition and reduced physical activity and sleep quality when they are taking modulator therapy compared to a healthy group.

The aims of this study are:

1. Determine the aerobic exercise function and mechanisms underlying this in people with CF stable on ETI and whether this is different to healthy age- and sex-matched controls;
2. Determine the peripheral muscle function in people with CF stable on ETI and whether this is different to healthy age- and sex-matched controls;
3. Determine the functional exercise capacity in people with CF stable on ETI and whether this is different to healthy age- and sex-matched controls;
4. Determine the micro- and macrovascular endothelial function in people with CF stable on ETI and whether this is different to healthy age- and sex-matched controls;
5. Determine body composition in people with CF stable on ETI and whether this is different to healthy age- and sex-matched controls;
6. Determine the physical activity levels and sleep duration and quality in people with CF stable on ETI and whether this is different to healthy age- and sex-matched controls

This study will recruit 50 people with CF and 50 healthy age- and sex-matched control participants who are older than 10 years of age. It will ask them to attend the University of Portsmouth for 2 visits. The first visit will last ~3 hours. During this time they will undergo measures on blood vessel function and aerobic exercise function. The second visit will last ~2 hours. During this time they will undergo a body composition scan and a series of muscle function test. At home, participants will wear an accelerometer for 7 days and complete a series of questionnaires.

ELIGIBILITY:
Inclusion criteria for participants with cystic fibrosis:

* Stable on the modulator therapy, Kaftrio®
* Males and females ≥ 10 years of age
* CF diagnosis based on clinical features, supported by a history of an abnormal sweat test (sweat chloride > 60 mmol·L-1 > 100 mg sweat), where possible, diagnostic genotyping would also be desired
* Can clearly state that they are not pregnant
* No contraindications to performing exercise
* Can understand and cooperate with the study protocol
* No increase in symptoms or weight loss in the preceding 2 weeks

Inclusion criteria for healthy control participants:

* Healthy males and females who are age- and sex-matched to the enrolled individuals with CF
* Can clearly state that they are not pregnant
* No clinical diagnosis of a chronic disease
* Can understand and cooperate with the study protocol
* No contraindications to performing exhaustive exercise

Exclusion criteria for participants with cystic fibrosis:

* Any non-pulmonary conditions that may impair exercise ability, such as musculoskeletal disorders and cardiovascular disease.
* Unstable co-morbid asthma (daily pulmonary function variability of >20%)
* Is pregnant during the initial screening process
* Unable to understand or cooperate with the study protocol due to learning difficulties or otherwise
* Not of a suitable age for testing
* Is a smoker or inhales any other substances
* Are taking vasoactive medications

Exclusion criteria for healthy control participants:

* Any pulmonary, metabolic or cardiovascular conditions
* Any other diagnosed disease
* Any non-pulmonary conditions that may impair exercise ability, such as musculoskeletal disorders and cardiovascular disease
* Is pregnant during the initial screening procedure
* Presents with co-morbidities to performing exhaustive exercise
* Is a smoker or inhales any other substance
* Unable to understand or cooperate with the study protocol due to learning difficulties or otherwise
* Not an age- or sex-match for the CF group
* Are taking vasoactive medications

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from adult and paediatric CF outpatient clinics within the Southampton CF network.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen uptake | Day 1 - baseline
  Between group differences in maximal oxygen uptake derived from a maximal cardiopulmonary exercise testing on a cycle ergometer

SECONDARY OUTCOMES:
Peak minute ventilation | Day 1 - baseline
  Between group differences in peak minute ventilation derived from a maximal cardiopulmonary exercise test on a cycle ergometer
Oxygen uptake at the gas exchange threshold | Day 1 - baseline
  Between group differences in oxygen uptake at the gas exchange threshold derived from a maximal cardiopulmonary exercise test on a cycle ergometer
Peak power output | Day 1 - baseline
  Between group differences in peak power output derived from a maximal cardiopulmonary exercise test on a cycle ergometer
Time to exhaustion | Day 1 - baseline
  Between group differences in time to exhaustion derived from a maximal cardiopulmonary exercise test on a cycle ergometer
Heart rate | Day 1 - baseline
  Between group differences in heart rate derived from a maximal cardiopulmonary exercise test on a cycle ergometer
Near-infrared spectroscopy derived deoxygenated [haemoglobin + myoglobin] | Day 1 - baseline
  Between group differences in dynamics of near-infrared spectroscopy derived deoxygenated [haemoglobin + myoglobin]
Cardiac output | Day 1 - baseline
  Between group differences in dynamics of non-invasive thoracic impedance cardiography
Stroke volume index | Day 1 - baseline
  Between group differences in dynamics of non-invasive thoracic impedance cardiography
Forced Expiratory Volume in the 1st second (% predicted) | Day 1 - baseline
  Between group differences in Forced Expiratory Volume in the 1st second measured using flow-volume loop spirometry
Forced Vital Capacity (%predicted) | Day 1 - baseline
  Between group differences in Forced Vital Capacity measured using flow-volume loop spirometry
Total minutes of physical activity (light, moderate, moderate to vigorous physical activity) | Physical activity will be measured continuously for 7 days
  Between group differences in physical activity assessed via wrist-worn accelerometery
Sleep efficiency (time in bed + time asleep) | Sleep efficiency will be measured continuously for 7 days
  Between group differences in sleep efficiency assessed via wrist-worn accelerometery
Acetylcholine iontophoresis | Day 1 - baseline
  Between group differences in acetylcholine iontophoresis measure of microvascular function
Insulin iontophoresis | Day 1 - baseline
  Between group differences in insulin iontophoresis measure of microvascular function
Percentage change in brachial artery diameter taken from the Flow Mediated Dilation assessment | Day 1 - baseline
  Between group differences in Flow Mediated Dilation assessment derived from baseline brachial artery diameter and peak brachial artery diameter from flow mediated dilation measure of macrovascular function
Maximum quadricep strength | Day 2 - baseline
  Derived from a maximal voluntary contraction
Quadricep fatigability index | Day 2 - baseline
  Derived from change in maximal voluntary contraction
Handgrip strength | Day 2 - baseline
  Between group difference in handgrip strength
Sit to stand repetitions per minute | Day 2 - baseline
  Between group difference in sit to stand repetitions per minute
Body composition (total fat-free mass and total fat mass) | Day 2 - baseline
  Derived from dual-energy X-ray absorptiometry
Habitual activity estimation scale | Day 2 - baseline
  Between group difference in habitual activity estimation scale - answers are varied and require numerical values, percentages and/or multiple choice questions
Cystic fibrosis questionnaire revised | Day 2 - baseline
  Between group difference in health related quality of life on a 0 - 100 scale with higher scores indicating better health related quality of life
The Pittsburgh Sleep Quality Index | Day 2 - baseline
  Between group differences in the Pittsburgh Sleep Quality Index on a 0 - 21 scale with higher scores indicating worse sleep quality
Perceived exertion (breathing effort, chest tightness, throat narrowing, perceived exertion) | Day 1 - baseline
  Between group differences in perceived exertion using the Dalhousie Dyspnoea and Perceived Exertion Scales during a maximal cardiopulmonary exercise testing on a cycle ergometer on a 1 - 7 scale with a higher value indicating a worse perceived exertion

CONTACTS AND LOCATIONS:
Locations (1):
- University of Portsmouth, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No